CLINICAL TRIAL: NCT03168334
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2 Arm, Parallel Group Study Comparing the Safety and Efficacy of IDP-123 Lotion and IDP-123 Vehicle Lotion in the Treatment of Acne Vulgaris
Brief Title: A Phase 3, Vehicle-controlled Efficacy and Safety Study of IDP-123 Lotion in the Treatment of Acne Vulgaris (302)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-123A-302
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-123 Lotion (Experimental): Tazarotene 0.045% Lotion
  Interventions: Drug: IDP-123 Lotion
- IDP-123 Vehicle Lotion (Placebo Comparator): Vehicle Lotion
  Interventions: Drug: IDP-123 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-123 Lotion — Tazarotene 0.045% Lotion
  Other Names: IDP-123
  Arms: IDP-123 Lotion
Drug: IDP-123 Vehicle Lotion — Vehicle Lotion
  Other Names: Vehicle
  Arms: IDP-123 Vehicle Lotion

SUMMARY:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, efficacy, and tolerability of IDP-123 Lotion in comparison with IDP-123 Vehicle Lotion.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, efficacy, and tolerability of IDP-123 Lotion and IDP-123 Vehicle Lotion. To be eligible for the study subjects must be at least 9 years of age and have a clinical diagnosis of moderate to severe acne.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 9 years of age and older;
2. Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit);
3. Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity assessment at the baseline visit;
4. Subjects with facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 20 but no more than 50;
5. Subjects with facial acne non-inflammatory lesion (open and closed comedones) count no less than 25 but no more than 100;
6. Subjects with two or fewer facial nodules

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study;
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis, dermatitis, eczema;
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
4. Subjects with a facial beard or mustache that could interfere with the study assessments;
5. Subjects with more than two (2) facial nodules;
6. Evidence or history of cosmetic-related acne

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (45):
- United States (41):
  - Valeant Site 41, Mobile, Alabama
  - Valeant Site 22, Rogers, Arkansas
  - Valeant Site 34, Carlsbad, California
  - Valeant Site 12, Fremont, California
  - Valeant Site 06, San Diego, California
  - Valeant Site 13, San Diego, California
  - Valeant Site 31, San Diego, California
  - Valeant Site 36, Santa Ana, California
  - Valeant Site 25, Denver, Colorado
  - Valeant Site 05, Boynton Beach, Florida
  - Valeant Site 29, Clearwater, Florida
  - Valeant Site 38, Jupiter, Florida
  - Valeant Site 02, Miami, Florida
  - Valeant Site 26, West Palm Beach, Florida
  - Valeant Site 44, Snellville, Georgia
  - Valeant Site 32, Louisville, Kentucky
  - Valeant Site 19, Rockville, Maryland
  - Valeant Site 08, Bay City, Michigan
  - Valeant Site 30, Clarkston, Michigan
  - Valeant Site 37, Clinton Township, Michigan
  - Valeant Site 20, Fort Gratiot, Michigan
  - Valeant Site 24, Fridley, Minnesota
  - Valeant Site 03, Morristown, New Jersey
  - Valeant Site 42, Albuquerque, New Mexico
  - Valeant Site 10, New York, New York
  - Valeant Site 43, Rochester, New York
  - Valeant Site 33, Stony Brook, New York
  - Valeant Site 11, Oklahoma City, Oklahoma
  - Valeant Site 28, Broomall, Pennsylvania
  - Valeant Site 16, Warwick, Rhode Island
  - Valeant Site 18, Knoxville, Tennessee
  - Valeant Site 14, Murfreesboro, Tennessee
  - Valeant Site 23, College Station, Texas
  - Valeant Site 07, Dallas, Texas
  - Valeant Site 27, Pflugerville, Texas
  - Valeant Site 04, San Antonio, Texas
  - Valeant Site 39, Sugar Land, Texas
  - Valeant Site 09, Layton, Utah
  - Valeant Site 15, West Jordan, Utah
  - Valeant Site 21, Charlottesville, Virginia
  - Valeant Site 35, Walla Walla, Washington
- Canada (4):
  - Valeant Site 01, Surrey, British Columbia
  - Valeant Site 45, Winnipeg, Manitoba
  - Valeant Site 40, Windsor, Ontario
  - Valeant Site 17, Saint-Jérôme, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IDP-123 Lotion: IDP-123 (Tazarotene 0.045%) Lotion
- Vehicle Lotion: IDP-123 Vehicle Lotion
Period: Overall Study
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Started | 397 | 404
Completed | 345 | 366
Not Completed | 52 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-123 Lotion | Vehicle Lotion | Total
Number analyzed (Participants) | 397 | 404 | 801
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (6.48) | 20.5 (6.81) | 20.3 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 262 | 513
  Male | 146 | 142 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 27 | 23 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 49 | 54 | 103
  White | 298 | 303 | 601
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 9 | 12 | 21
Lesion counts [Mean (Standard Deviation); unit: lesions] — For noninflammatory facial lesions, open comedones (blackheads) and closed comedones (whiteheads) were recorded as a single count. For inflammatory facial lesions, papules (solid, elevated lesion less than 5 mm) and pustules (elevated lesion containing pus less than 5 mm) were recorded as a single count, while nodular lesions (palpable subcutaneous lesion greater than 5 mm) were counted and recorded separately.
  lesions
    Non-inflammatory lesions | 41.8 (17.87) | 40.6 (16.31) | 41.2 (17.10)
    Inflammatory lesions | 28.0 (7.32) | 27.9 (7.10) | 28.0 (7.21)
Evaluator's Global Severity Score [Count of Participants; unit: Participants] — Evaluator's Global Severity Score (EGSS) was determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations were scored on a scale of 0-4, with 0 being clear and 4 being severe.
  Participants
    Moderate | 358 | 357 | 715
    Severe | 39 | 47 | 86

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Lesion Counts at Week 12
Description: For noninflammatory facial lesions, open comedones (blackheads) and closed comedones (whiteheads) were recorded as a single count. For inflammatory facial lesions, papules (solid, elevated lesion less than 5 mm) and pustules (elevated lesion containing pus less than 5 mm) were recorded as a single count, while nodular lesions (palpable subcutaneous lesion greater than 5 mm) were counted and recorded separately.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 397 | 404
lesion counts
  Non-inflammatory lesions | -24.6 (15.33) | -16.6 (15.48)
  Inflammatory lesions | -16.7 (9.49) | -13.4 (9.37)

2. Primary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS) and Had an EGSS at Week 12 That Equated to "Clear" or "Almost Clear"
Description: Evaluator's Global Severity Score (EGSS) was determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations were scored on a scale of 0-4, with 0 being clear and 4 being severe.
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 397 | 404
percentage of participants | 29.6 | 17.3

3. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 397 | 404
percentage change
  Non-inflammatory lesions | -60.00 (34.680) | -41.58 (35.239)
  Inflammatory lesions | -59.50 (33.382) | -48.95 (32.898)

4. Secondary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 397 | 404
percentage of participants | 34.5 | 20.9

5. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 397 | 404
percentage change
  Non-inflammatory lesions | -48.45 (36.497) | -30.92 (36.772)
  Inflammatory lesions | -50.38 (32.917) | -41.66 (32.874)

6. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 397 | 404
percentage change
  Non-inflammatory lesions | -35.03 (32.776) | -24.12 (33.040)
  Inflammatory lesions | -32.31 (32.906) | -31.55 (32.954)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety population included all participants who received at least one confirmed dose of study drug and had at least one post-baseline safety assessment. There were 10 participants in the IDP-123 Lotion and 12 participants in the IDP-123 Vehicle Lotion group who did not have any post- baseline safety assessment.
Arm/Group | IDP-123 Lotion | Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/387 | 0/392
Serious Adverse Events (participants affected / at risk) | 1/387 | 1/392
Other Adverse Events (participants affected / at risk) | 43/387 | 17/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-123 Lotion (N=387) | Vehicle Lotion (N=392)
Abortion induced (Surgical and medical procedures) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-123 Lotion (N=387) | Vehicle Lotion (N=392)
Application Site Pain (General disorders) | 23 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 20 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT03168334/Prot_SAP_000.pdf